CLINICAL TRIAL: NCT05004428
Title: Chronic Kidney Disease in Type 2 Diabetes Mellitus
Brief Title: A Study to Learn More About Chronic Kidney Disease (CKD) in Patients With Type 2 Diabetes Mellitus (T2DM)
Acronym: CKD-T2DM
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21510
Record Dates: First submitted 2021-07-14; First posted 2021-08-13 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Disease
Keywords: Cardiovascular Diseases; Kidney Diseases; Renal Insufficiency, Chronic; Diabetes Mellitus , Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Cardiovascular Diseases; Kidney Diseases; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 Diabetes Mellitus patients with Chronic Kidney Disease: Canadian patients with type 2 diabetes mellitus data will be collected retrospectively.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Retrospective population-based study utilizing administrative data without any intervention.

SUMMARY:
In this observational study, data from the recent past of patients with type 2 diabetes mellitus and chronic kidney disease will be studied.

Type 2 diabetes mellitus (T2DM) is a condition in which the body does not make enough of a hormone called insulin or does not use insulin well. This results in high blood sugar levels. About half of people with T2DM also have a condition called chronic kidney disease (CKD). In people with CKD, the kidneys' ability to work as how it should decreases over time.

In this study, researchers want to learn more about the CKD in T2DM patients in Alberta, Canada. This will help them to know the chances to improve the care of these patients.

The researchers will look at the health information from adult men and women in Alberta who were diagnosed with T2DM before 2018 and visited a doctor to have check-ups in 2018. They will find out about how many of these people had CKD and how severe their CKD was. The researchers will collect data about the age and gender of these patients, how long they had T2DM and if they had other related medical problems. The researchers will also learn how these patients were treated based on their kidney condition and how much money was spent on these treatments.

This study will collect information from the health records of about 270,000 patients with T2DM who were living in Alberta, Canada. This information will come from the Alberta Kidney Disease Network (AKDN) database. Besides this data collection, no further tests or examinations are planned in this study.

ELIGIBILITY:
Inclusion Criteria:

* A cohort of adults (18 years and older) with Type 2 Diabetes Mellitus (T2DM) who resided in Alberta on the index date (December 31, 2018) and were registered with Alberta Health will be included. All Alberta residents are eligible for Alberta Health Insurance Plan coverage and over 99% participate.

Exclusion Criteria:

* Patients with type 1 DM (T1DM) (International Classification of Diseases, Ninth Revision [ICD-9] code: 250.x1 and 250.x3) in any of their previous records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients medical history data from Alberta Kidney Disease Network (AKDN) with Type 2 diabetes by chronic kidney disease (CKD) stage and by rate of CKD progression will be collected retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 336376 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Type 2 Diabetes Mellitus (T2DM) patients with Chronic Kidney Disease (CKD) in database. | Baseline
  Percentage of T2DM patients with CKD as per hemoglobin A1C, and stage of CKD as defined by a) baseline Kidney Disease: Improving Global Outcomes (KDIGO) guidelines CKD category, and b) eGFR ≥25 to <75 mL/min/1.73 m2 and ACR ≥30 to ≤5,000 mg/g.

SECONDARY OUTCOMES:
Descriptive analyses of clinical characteristics of patients in database. | Baseline
  Duration of diabetes, comorbities and slope of eGFR
Descriptive analyses of demographic data. | Baseline
  Age, sex, urban or rural residence.
Rate of decline in estimated glomerular filtration rate (eGFR) | Retrospectively 3 years
Number of patients with CKD dispensed the medication or therapeutic class over a 1-year time period | from January 1, 2018 to December 31, 2018
The proportion of patients with CKD that experience a health outcome of interest over a 1-year time period | from January 1, 2018 to December 31, 2018
Health care resource utilization among patients | from January 1, 2018 to December 31, 2018
Annual average costs among patients | from January 1, 2018 to December 31, 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Canada

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/